CLINICAL TRIAL: NCT02654041
Title: Phase II, Open-label, Prospective, Single-arm, Single-center Study of Induction of Hypothyroxinemia Adjunct to Conventional Therapies in GBM Patients
Brief Title: Study of Induction of Hypothyroxinemia Adjunct to Conventional Therapies in GBM Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug manufacturer no longer could supply for study
Sponsor: Musli Thyropeutics Ltd. (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MusliGBM002
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2016-11

CONDITIONS: Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypothyroxinemia induced patients (Experimental): Combined T3 and Methimazole treatment will be administered. This experimental treatment will be administered adjunct to standard oncological treatment for newly-diagnosed GBM patients e.g. radiation followed by Temozolomide.
  Interventions: Drug: Combined T3 and Methimazole treatment

INTERVENTIONS:
Drug: Combined T3 and Methimazole treatment — Oral administration of T3 and Methimazole

SUMMARY:
The objective of the study is to assess the safety and efficacy of treatment with hypothyroxinemia adjunct to conventional therapies in GBM patients.

DETAILED DESCRIPTION:
Since T4 (thyroxine) is a potent growth factor in numerous cancer types, the interventional approach will be to achieve thyroxine deprivation (hypothyroxinemia).This can be achieved by using a dual approach: T3 and methimazole to provide longer term inhibition of thyroid hormone synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GBM, histologically or cytologically confirmed.
* Newly-diagnosed subjects prior to beginning first-line conventional therapy.
* Male or female subjects 18 years of age or older.
* Ability to understand and willingness to sign a written informed consent document.
* Ability and consent to comply with completion of a patient diary.
* Subjects must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) with conventional techniques or as ≥10 mm (≥1 cm) with spiral CT scan, MRI, or calipers by clinical exam.
* Allowable type and amount of prior therapy and medication
* ECOG performance status ≤2 (KPS ≥60%, see Appendix A).
* Life expectancy of greater than 6 months
* Subjects must have adequate bone marrow, liver and renal function as assessed by the following laboratory requirements conducted within 7 days of starting to study treatment:
* Total bilirubin < 1.5 x the upper limit of normal (ULN).
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) < 2.5 xULN (< 5 x ULN for subjects with liver involvement of their cancer).
* Alkaline phosphatase limit < 2.5 x ULN (<5 x ULN for subjects with liver involvement of their cancer)
* Serum creatinine < 1.5 x the ULN. Glomerular filtration rate (GFR) ≥ 30 ml/min/1.73 m2 according to the MDRD (Modified diet in renal disease) abbreviated formula.
* INR/PTT < 1.5 x ULN.
* Platelet count > 100000 /mm3, Hemoglobin (Hb) > 9 g/dl, Absolute neutrophil count (ANC) > 1500/mm3
* No significant abnormalities in serum hematology, serum chemistry and serum inflammatory / immunogenic markers according to the Principal Investigator's judgment.
* No significant abnormalities in urinalysis according to the Principal Investigator's judgment, taking into considerations the potential effects of the tumor.
* No significant abnormalities in ECG per investigator judgment.
* Non-pregnant, non-lactating female subjects.
* Women of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study.

Exclusion Criteria:

* Patients unable to swallow oral medications.
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Patients who are receiving any other investigational agents or participating in another interventional clinical trial within 30 days prior to baseline visit (patients participating in other observational trials are allowed to be enrolled in this study).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to anti-thyroid agent (such as methimazole or PTU) or Cytomel®, or other agents used in study.
* Current or prior (within the last 60 days prior to screening visit) use of any medication or substance that have the potential to affect the activity or pharmacokinetics of the study agents (please refer to package inserts of study drugs).
* Specific none-allowable type and amount of prior therapy and medication
* Clinically significant concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active connective tissue disorders, such as lupus or scleroderma, human immunodeficiency virus or psychiatric illness/social situations that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study and would limit compliance with study requirements.
* History of organ allograft.
* Non-healing wound, ulcer, or bone fracture.
* Renal failure requiring hemo-or peritoneal dialysis.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
* Evidence of uncontrolled hypertension (systolic blood pressure of >150 mm Hg, and/or diastolic blood pressure of >100 mm Hg) (at any time) when taken 3 times on the same arm with the subject in the supine position.
* Evidence of alcohol abuse or history of alcohol abuse or illegal and/or legally prescribed drugs.
* Inability to attend scheduled clinic visits and/or comply with the study protocol.
* Any other factor that, in the opinion of the investigator, would prevent the patient from complying with the requirements of the protocol.
* Any prior abnormalities related to the thyroid and /or intake of thyroid related drugs (e.g Eltroxin) in the 3 months prior to the study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Response rate at 6 months (6 months PFS) | 32 weeks
  The primary outcome measure of the study is the ratio of patients who complete their 6-month course of chemotherapy given the IP adjunct treatment. Each patient is treated up to 6 weeks until their FT4 target is reached at which time they enter a 26 week (6 month) treatment phase during which they receive chemotherapy as per common protocol with the IP as adjunct treatment. Patients will be monitored for disease progression as per common oncological protocol (e.g. every 2 months) and those who show progression will be deemed failures. Patients with no disease progression (or partial or complete remission) at the end of the 6 month period will be considered success.

SECONDARY OUTCOMES:
Response rate at 2 months (2 months PFS) | 14 weeks
  As a secondary outcome we will measure 2 month progression free survival as measured by RANO.
Response rate at 4 months (4 months PFS) | 23 weeks
  As a secondary outcome we will measure 4 month progression free survival as measured by RANO.
Time to disease progression or cancer-related death | 32 weeks
Safety endpoint evaluation | 32 weeks
  Patients will be monitored throughout the study period for any Hypothyroxinemia treatment related safety issues including serious adverse events, any adverse events, vital signs, lab assessment, physical examination and lung function.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah T Blumenthal, MD, Principal Investigator — Tel-Aviv Medical Center, Israel
Locations (1):
- Tel-Aviv Medical Center, Israel, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided